CLINICAL TRIAL: NCT06852729
Title: Effect of Induced Trunk Extensors Fatigue on Balance and Lumbar Position Sense in Adolescents
Acronym: LPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AHMED GAMAL ABD EL-NASSER ALI, Principal investigator ahmed gamal abd el-nasser ali, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005624
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Adolescent
Keywords: induced trunk extensor fatigue; balance; Lumbar Position Sense

STUDY DESIGN:
Intervention Model Description: Biering-sorenson protocol will be applied to induce back muscle fatigue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biering-sorenson protocol (Experimental): Biering-Sorensen protocol will be used to induce back muscle fatigue, and a marked decrease in the maximum force in trunk extension
  Interventions: Other: Biering-sorenson protocol

INTERVENTIONS:
Other: Biering-sorenson protocol — * Students shouldn't perform any vigorous activity a day before assessment.
  * Frist, therapist will request from each participant to watch videos to understand how the test should be applied.
  * The starting position will be a half prone lying on a plinth with the superior edge of the iliac crest horizontal at the edge of the plinth and the arms crossed over the chest.
  * The participant should keep the unsupported upper part of the body.
  * The lower limbs will strategically be stabilized with straps.
  * The participant will be asked to maintain the upper body in a horizontal position and the timer started.
  * The test ends if the participant can maintain the previous position for 4 minutes (240 seconds) or can no longer maintain the set position before 4 minutes elapses. The stop time is recorded.
  * There is considerable range of mean fatigue times reported for the Biering-Sørensen test in the literature ranging from 84s to 180s in healthy males.

SUMMARY:
this study will be conducted to investigate the effect of trunk extensors induced fatigue on balance and lumber position sense in adolescents

DETAILED DESCRIPTION:
Fatigue can be defined as, decrease in the power generation capacity of the muscles from the beginning of the movement due to internal homeostasis breakdown caused by an increase in energy production demanded by an external stimulus that lead to general decrease in physical performance related to a rise within the real/perceived difficulty of a task or exercise, as well as the inability of the muscles to keep up with the specified level of strength during exercises. Either Adolescents spending long time using smartphone, they are more likely to have their spine in an incorrect posture causing damage to the surrounding skeletal structures as well as to ligaments which affect the proprioception input of the spine. Muscle fatigue is an important condition that impairs sensorimotor integration, proprioception, and thus postural control. Muscle fibers and Golgi tendon organ activity decrease with fatigue, resulting in changes in joint proprioception and afferent output from joint and muscle receptors. Fatigue of postural muscles such as lumbar extensor and abdominal muscles impairs postural control and may form the basis for injuries. Fatigue can also impair the proprioceptive and kinesthetic properties of the joints. this study aims to investigate how the trunk extensor muscles respond to a fatigue inducing exercise, especially concerning balance and trunk lumbar position sense for understanding and preventing musculoskeletal injury and lowering risk in health adolescents in primary care and to contribute to preventive rehabilitation. Sixty-eight normal adolescent boys will participate in this study

ELIGIBILITY:
Inclusion Criteria:

* Only boys will be included.
* Their age will range from 16 to 18 years old.
* Never trained any specific sport before.
* They have a normal body mass index (BMI) between 16.4 to 24.8 kg/m2 according to
* No history of low back (pain intensity 0-1 cm) according to 10 cm visual analog scale (VAS)
* Physical fitness of all participants will be (minimally active) according to International Physical Activity Questionnaire- Short Form (IPAQ-SF)

Exclusion Criteria:

* Visual or hearing defects.
* Congenital abnormalities.
* Musculoskeletal abnormalities.
* Recent trauma.
* Cardiac and respiratory problems.
* Smoker participant.
* Low back pain.

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
balance | up to thirty minutes
  Assessment of balance will be done using the biodex balance system
joint position error | up to thirty minutes
  Inclinometer will be used to assess lumbar joint position error